CLINICAL TRIAL: NCT00345163
Title: A Phase II, Multicenter, Randomized, Non-Comparative Clinical Trial to Evaluate the Efficacy and Safety of Bevacizumab Alone or in Combination With Irinotecan for Treatment of Glioblastoma Multiforme in First or Second Relapse
Brief Title: A Study to Evaluate Bevacizumab Alone or in Combination With Irinotecan for Treatment of Glioblastoma Multiforme (BRAIN)
Acronym: BRAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVF3708g
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Glioblastoma
Keywords: Glioblastoma Multiforme; Avastin; Brain Cancer; GBM
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Bevacizumab; Irinotecan

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab
- 2 (Experimental)
  Interventions: Drug: bevacizumab; Drug: irinotecan

INTERVENTIONS:
Drug: bevacizumab — Intravenous repeating dose
Drug: irinotecan — Intravenous repeating dose
  Arms: 2

SUMMARY:
This is a Phase II, open-label, multicenter, randomized, non comparative study consisting of two concurrent single-arms. Approximately 160 subjects will be randomized in a 1:1 ratio to Arm 1 (bevacizumab alone) or Arm 2 (bevacizumab + irinotecan).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥ 18 years
* Histologically confirmed GBM in first or second relapse
* Radiographic demonstration of disease progression following prior therapy
* Bi-dimensionally measurable disease with a minimum measurement of 1 cm (10 mm) in one diameter on MRI performed within 14 days prior to first treatment (Day 0)
* An interval of ≥ 4 weeks since prior surgical resection
* Prior standard radiation for GBM
* Prior chemotherapy: first-relapse subjects
* Prior chemotherapy: second-relapse subjects
* Recovery from the effects of prior therapy, including the following: 4 weeks from cytotoxic agents (except 6 weeks from nitrosoureas, 3 weeks from procarbazine, 2 weeks from vincristine); 4 weeks from any investigational agent; 1 week from non-cytotoxic agents; 8 weeks from radiotherapy to minimize the potential for MRI changes related to radiation necrosis that might be misdiagnosed as progression of disease, or 4 weeks if a new lesion, relative to the pre-radiation MRI, develops that is outside the primary radiation field
* Prior therapy with gamma knife or other focal high-dose radiation is allowed but the subject must have subsequent histologic documentation of recurrence, unless the recurrence is a new lesion outside the irradiated field
* Karnofsky performance status ≥ 70
* Life expectancy > 12 weeks
* Use of an effective means of contraception in males and in females of childbearing potential
* Ability to comply with study and follow-up procedures

Exclusion Criteria:

* Prior treatment with irinotecan, bevacizumab, or another VEGF or VEGFR-targeted agent
* Prior treatment with prolifeprospan 20 with carmustine wafer
* Prior intracerebral agents
* Need for urgent palliative intervention for primary disease (e.g., impending herniation)
* Evidence of recent hemorrhage on baseline MRI of the brain with the following exceptions: Presence of hemosiderin; Resolving hemorrhagic changes related to surgery; Presence of punctate hemorrhage in the tumor
* Received more than two treatment regimens for Grade III and/or Grade IV glioma
* Blood pressure of > 150 mmHg systolic and > 100 mmHg diastolic
* History of hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater CHF
* History of myocardial infarction or unstable angina within 6 months prior to Day 0
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis within 6 months prior to Day 0
* Evidence of bleeding diathesis or coagulopathy
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* History of intracerebral abscess within 6 months prior to Day 0
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures (excluding placement of a vascular access device), stereotactic biopsy, fine needle aspirations, or core biopsies within 7 days prior to Day 0
* Serious non-healing wound, ulcer, or bone fracture
* Pregnancy (positive pregnancy test) or lactation
* Known hypersensitivity to any component of bevacizumab
* History of any other malignancy within 5 years (except non-melanoma skin cancer or carcinoma in situ of the cervix)
* Pregnant or nursing females
* Unstable systemic disease, including active infection, uncontrolled hypertension, or serious cardiac arrhythmia requiring medication
* Subjects unable to undergo an MRI with contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Objective response, as determined by the independent review facility (IRF) | Complete response or partial response, determined on two consecutive assessments ≥4 weeks apart
Progression-free survival, as determined by the IRF | 6 months

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | Length of patient on study
Duration of objective response, as determined by the IRF | Complete or partial response determined on two consecutive assessments ≥4 weeks apart
Overall survival | Time from randomization to death

CONTACTS AND LOCATIONS:
Overall Officials: Jane Huang, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Result] Friedman HS, Prados MD, Wen PY, Mikkelsen T, Schiff D, Abrey LE, Yung WK, Paleologos N, Nicholas MK, Jensen R, Vredenburgh J, Huang J, Zheng M, Cloughesy T. Bevacizumab alone and in combination with irinotecan in recurrent glioblastoma. J Clin Oncol. 2009 Oct 1;27(28):4733-40. doi: 10.1200/JCO.2008.19.8721. Epub 2009 Aug 31. PMID 19720927
- [Derived] Ellingson BM, Hagiwara A, Morris CJ, Cho NS, Oshima S, Sanvito F, Oughourlian TC, Telesca D, Raymond C, Abrey LE, Garcia J, Aftab DT, Hessel C, Rachmilewitz Minei T, Harats D, Nathanson DA, Wen PY, Cloughesy TF. Depth of Radiographic Response and Time to Tumor Regrowth Predicts Overall Survival Following Anti-VEGF Therapy in Recurrent Glioblastoma. Clin Cancer Res. 2023 Oct 13;29(20):4186-4195. doi: 10.1158/1078-0432.CCR-23-1235. PMID 37540556
- [Derived] Ellingson BM, Harris RJ, Woodworth DC, Leu K, Zaw O, Mason WP, Sahebjam S, Abrey LE, Aftab DT, Schwab GM, Hessel C, Lai A, Nghiemphu PL, Pope WB, Wen PY, Cloughesy TF. Baseline pretreatment contrast enhancing tumor volume including central necrosis is a prognostic factor in recurrent glioblastoma: evidence from single and multicenter trials. Neuro Oncol. 2017 Jan;19(1):89-98. doi: 10.1093/neuonc/now187. Epub 2016 Aug 31. PMID 27580889
- [Derived] Ellingson BM, Kim HJ, Woodworth DC, Pope WB, Cloughesy JN, Harris RJ, Lai A, Nghiemphu PL, Cloughesy TF. Recurrent glioblastoma treated with bevacizumab: contrast-enhanced T1-weighted subtraction maps improve tumor delineation and aid prediction of survival in a multicenter clinical trial. Radiology. 2014 Apr;271(1):200-10. doi: 10.1148/radiol.13131305. Epub 2013 Nov 27. PMID 24475840